CLINICAL TRIAL: NCT02467348
Title: To Study the Incidence And Outcome Of Paracentesis Induced Circulatory Dysfunction In Acute-On-Chronic Liver Failure Undergoing Less Than 5 Litres Of Ascitic Fluid Tap With Or Without Albumin Infusion.
Brief Title: Incidence And Outcome Of Paracentesis Induced Circulatory Dysfunction In Acute-On-Chronic Liver Failure.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institute of Liver and Biliary Sciences, India (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ILBS-ACLF and Cirrhosis-01
Record Dates: First submitted 2015-06-04; First posted 2015-06-10 (Estimated); Last update posted 2017-11-28 (Actual); Status verified 2017-01

CONDITIONS: Acute on Chronic Liver Failure
MeSH Terms: conditions — Acute-On-Chronic Liver Failure | interventions — Albumins

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Albumin (Experimental): MVP (Modest Volume Paracentesis) of less than 5 litres with intravenous albumin at a dose 8 gms/l of ascitic fluid.
  Interventions: Drug: Albumin; Drug: Ascitic fluid
- No Albumin (Active Comparator): MVP (Modest Volume Paracentesis) of less than 5 litres without albumin.
  Interventions: Drug: Ascitic fluid

INTERVENTIONS:
Drug: Albumin — Intravenous albumin 8 gms/L of ascitic fluid
  Arms: Albumin
Drug: Ascitic fluid

SUMMARY:
All consecutive patients admitted in ILBS from MAY 2015 to DECEMBER 2016.ACLF (Acute on chronic Liver Failure). ACLF will be randomize into

Group 1: MVP (Modest Volume Paracentesis) OF Less than 5 liters with IV albumin at a dose 8 gms/L of ascitic fluid

Group 2: MVP (Modest Volume Paracentesis) of Less than 5 liters without albumin

ELIGIBILITY:
Inclusion Criteria:

1. All patients with acute hepatic insult manifesting as jaundice (Sr. Bil. ≥ 5 mg/dL) and coagulopathy (INR≥1.5), complicated within 4 weeks by ascites and/or encephalopathy in a patient with previously diagnosed or undiagnosed chronic liver disease (ACLF) admitted in the hospital.
2. All Cirrhotics decompensated with ascites admitted in the hospital.
3. Grade II/III ascites
4. Need for paracentesis.

Exclusion Criteria:

1. Age <12 or > 75 years
2. Hepatocellular carcinoma
3. Non cirrhotic ascites such as malignancy or tubercular peritonitis
4. Serum Cr >1.5mg%
5. Refractory septic shock
6. Grade III/IV hepatic encephalopathy
7. Abdominal wall cellulitis
8. Active variceal bleed
9. Respiratory, cardiac and renal failure
10. Refusal to participate in the study

Ages: 12 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2015-03-15 (Actual); Primary Completion 2017-01-31 (Actual); Study Completion 2017-01-31 (Actual)

PRIMARY OUTCOMES:
Total number of patients develop Circulatory Dysfunction because of paracentesis. | 1 Year

SECONDARY OUTCOMES:
Survival | 28 days
Total number of patients develop hepatorenal Syndrome. | 1 Year
Total number of patients develop hyponatremia. | 1 Year
Changes in aldosterone with volume of ascitic fluid tap | 1 Year
Changes in plasma renin activity | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Liver and Biliary Sciences, New Delhi, National Capital Territory of Delhi, India

REFERENCES:
- [Derived] Arora V, Vijayaraghavan R, Maiwall R, Sahney A, Thomas SS, Ali R, Jain P, Kumar G, Sarin SK. Paracentesis-Induced Circulatory Dysfunction With Modest-Volume Paracentesis Is Partly Ameliorated by Albumin Infusion in Acute-on-Chronic Liver Failure. Hepatology. 2020 Sep;72(3):1043-1055. doi: 10.1002/hep.31071. Epub 2020 Jul 9. PMID 31849085